CLINICAL TRIAL: NCT05714865
Title: Less Invasive Surfactant Administration in Nigeria
Brief Title: Implementing LISA Surfactant in Nigeria
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: BLES Biochemicals Inc. (Unknown)
Responsible Party: Principal Investigator, Osayame Ekhaguere, Assistant Professor of Pediatrics, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NHREC/01/01/2007-12/10/2022
Record Dates: First submitted 2022-12-28; First posted 2023-02-06 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Respiratory Distress Syndrome; Neonatal Death
MeSH Terms: conditions — Respiratory Distress Syndrome; Perinatal Death | interventions — Surface-Active Agents

STUDY DESIGN:
Intervention Model Description: Prospective cohort
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LISA Arm (Experimental): Eligible subjects who have respiratory distress syndrome (Anderson Silverman Score >4) managed on continuous positive airway pressure (CPAP) will receive surfactant via a thin catheter while on CPAP.
  Interventions: Drug: Surfactant

INTERVENTIONS:
Drug: Surfactant — Laryngoscopy is performed, and BLES® surfactant is administered through BLEScath™ (a thin catheter) into the trachea to a spontaneously breathing preterm infant with respiratory distress syndrome who is being managed on CPAP
  Other Names: BLES® Surfactant; BLEScath™; Less Invasive Surfactant Administration

SUMMARY:
Implement surfactant (BLES®) replacement therapy using the Less Invasive Surfactant Administration technique in six tertiary institutions in Nigeria and evaluate its impact on 72-hour neonatal mortality in premature infants born less than 2000 grams at birth.

DETAILED DESCRIPTION:
Background: In low- and middle-income countries (LMICs), respiratory distress syndrome (RDS) accounts for ~45% of all in-hospital neonatal mortality. Surfactant use is limited in LMICs, in part, due to the high cost, the lack of skill to perform laryngoscopy and tracheal intubation, and perhaps a perception that surfactant administration and mechanical ventilation must occur together. In LMICs, continuous positive airway pressure (CPAP) is often the highest mode of respiratory support available, and CPAP failure invariably means death. If Less Invasive Surfactant Administration (LISA) can reduce CPAP failure, as shown in high-income settings, it potentially can reduce prematurity-related neonatal mortality in LMICs. There are, however, no studies on how to safely implement LISA in LMICs. The LISA procedure is novel in LMICs; the procedure is not without risk (severe and minor), laryngoscopy is a difficult skill to acquire, master, and maintain, and the resource limitations in LMICs need consideration while implementing LISA.

Hypothesis: Compared to a historical control, introducing non-invasive surfactant administration through the less invasive surfactant administration (LISA) techniques will result in a relative risk reduction of all-cause 72-hour in-hospital mortality by at least 20%.

PICO Outline:

Population: Preterm infants </= 2 kg with respiratory distress defined by a Downes Respiratory Distress Score of >4, who are spontaneously breathing, and on CPAP.

Intervention: Surfactant administered through the less invasive surfactant administration (LISA), technique.

Comparator: A historical control of preterm babies </= 2 kg with respiratory distress defined by a Downes Respiratory Distress Score of >4, who are spontaneously breathing, and on CPAP.

Outcome measures:

Primary Outcome: 72-hour all-cause in-hospital mortality.

Secondary outcomes

* All-cause in-hospital mortality
* Change in respiratory distress score, pre- to -post interventions.

ELIGIBILITY:
Inclusion Criteria:

* Newborns with birth weight between 500-2000 grams (determined by birth weight or admission weight if birth weight is unavailable).
* ≤48 Hours old at recruitment.
* Spontaneously breathing but have clinical signs of respiratory distress (defined by Anderson Silverman Score (ASS) ≥4 (range 0-10)) and on CPAP.
* Admitted to the neonatal/newborn units (or special care nurseries).

Exclusion Criteria:

* Any newborn intubated before admission to the neonatal/newborn units.
* Any newborn infants with a significant congenital abnormality
* Any preterm infant considered nonviable by the managing clinician.

Ages: 1 Hour to 2 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 349 (Actual)
Dates: Start 2023-06-25 (Actual); Primary Completion 2025-03-30 (Actual); Study Completion 2025-03-30 (Actual)

PRIMARY OUTCOMES:
72-hour mortality | 72 hours of life
  All cause mortality with 72-hours of life

SECONDARY OUTCOMES:
In-hospital mortality | Through hospitalization, an average of 1 day to 10 weeks.
  All cause mortality during hospitalization
Difference in RDS score before and after the procedure. | 6 hours post procedure
  Change in Anderson Silverman RDS Score before and after intervention (range: 0 to 10)

CONTACTS AND LOCATIONS:
Overall Officials: Osayame A Ekhaguere, MBBS, MPH, Principal Investigator — Indiana University School of Medicine
Locations (6):
- Nigeria (6):
  - Federal Medical Center Asaba, Asaba, Delta
  - University of Benin Teaching Hospital, Benin City, Edo
  - National Hospital Abuja, Garki, FCT Abuja
  - Aminu Kano Teaching Hospital, Zaria, Kano State
  - Lagos University Teaching Hospital., Idi Araba, Lagos
  - University of Nigeria Teaching Hospital, Enugu

IPD SHARING:
Plan to Share IPD: No
On request and approval from local principal investigators and ethical approval committee